CLINICAL TRIAL: NCT05760378
Title: An Open, Randomized Phase III Study of Famitinib With Camrelizumab Plus Treatment of Physician's Choice (TPC) Versus Camrelizumab Plus TPC in The First-line Treatment of Immunomodulatory Locally Advanced or Metastatic Triple-negative Breast Cancer
Brief Title: Famitinib in Combination With Camrelizumab and TPC in The First-line Treatment of Immunomodulatory Locally Advanced or Metastatic TNBC.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCTOP-T-M02
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-06

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — famitinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Famitinib in Combination With Camrelizumab and TPC
  Interventions: Drug: Famitinib; Drug: Camrelizumab; Drug: nab-Palitaxel/Capecitabine/Eribulin Mesylate/Carboplatin
- B (Active Comparator): Combination With Camrelizumab and TPC
  Interventions: Drug: Camrelizumab; Drug: nab-Palitaxel/Capecitabine/Eribulin Mesylate/Carboplatin

INTERVENTIONS:
Drug: Famitinib — TKI
  Arms: A
Drug: Camrelizumab — PD1 inhibitor
Drug: nab-Palitaxel/Capecitabine/Eribulin Mesylate/Carboplatin — TPC

SUMMARY:
The study is being conducted to evaluate the Famitinib with Camrelizumab plus treatment of physician's choice (TPC) versus Camrelizumab plus TPC in Patients with Unresectable Locally Advanced or Metastatic Immunomodulatory Triple Negative Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0-1
* Expected lifetime of not less than three months
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Cancer stage: recurrent or metastatic breast cancer; Local recurrence be confirmed by the researchers could not be radical resection.
* Adequate hematologic and end-organ function, laboratory test results.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) • Patients had received no previous chemotherapy or targeted therapy for metastatic triple-negative breast cancer

Exclusion Criteria:

* Previous received anti-VEGFR small molecule tyrosine kinase inhibitors (e.g. famitinib, sorafenib, Sunitinib, regorafenib, etc.) for treatment of the patients .
* A history of bleeding, any serious bleeding events.
* Important blood vessels around tumors has been infringed and high risk of bleeding.
* Coagulant function abnormality
* artery/venous thromboembolism event
* History of autoimmune disease
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Uncontrolled pleural effusion and ascites • Known central nervous system (CNS) disease.
* Long-term unhealing wound or incomplete healing of fracture
* urine protein ≥2+ and 24h urine protein quantitative > 1 g.
* Pregnancy or lactation.
* Thyroid dysfunction.
* Peripheral neuropathy grade ≥2.
* People with high blood pressure;
* A history of unstable angina;
* New diagnosis of angina pectoris.
* Myocardial infarction incident .

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 1.5 years)
  time to progressive disease (according to RECIST1.1)

SECONDARY OUTCOMES:
ORR | max 6 months
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)
DoR | max 6 months
  Duration of Overall Response.The date of the first assessed PR/CR (according to RECIST 1.1) to the date of the first assessed tumor progression (according to RECIST 1.1) or death from any cause.
CBR | max 6 months
  The percentage of subjects with CR+PR+SD and last more than 24 weeks in all of the participants.
OS | approximately 3 years
  time to death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China